CLINICAL TRIAL: NCT06652971
Title: A Randomized, Open-label, Single-dose, Cross-over Phase 1 Study to Evaluate the Effect of Food on Pharmacokinetic Characteristics and Safety of CKD-379 in Healthy Adult Volunteers
Brief Title: A Clinical Trial to Evaluate the Food Effect of CKD-379
Acronym: CKD-379
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A125_06FDI2411
Record Dates: First submitted 2024-10-21; First posted 2024-10-22 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence 1 (Experimental): Period 1: A single oral dose of 1 tablet under fasting condition Period 2: A single oral dose of 1 tablet under fed condition
  Interventions: Drug: CKD-379
- Sequence 2 (Experimental): Period 1: A single oral dose of 1 tablet under fed condition Period 2: A single oral dose of 1 tablet under fasting condition
  Interventions: Drug: CKD-379

INTERVENTIONS:
Drug: CKD-379 — QD, PO

SUMMARY:
A clinical trial to evaluate the food effect of CKD-379

DETAILED DESCRIPTION:
A randomized, open-label, single-dose, cross-over phase 1 study to evaluate the effect of food on pharmacokinetic characteristics and safety of CKD-379 in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult aged 19 or older and 55 or younger at screening
2. Body mass index (BMI) of 18.0 kg/m2 or more and less than 30.0kg/m2 and Body weight ≥ 50kg
3. Those with systolic blood pressure ≤ 150 mmHg and ≥ 90 mmHg, diastolic blood pressure ≤ 100 mmHg and ≥ 50 mmHg
4. A person who has no clinically significant congenital or chronic diseases and has no pathological symptoms or findings as a result of medical examination
5. A person determined to be suitable for testing as a result of diagnostic tests and electrocardiogram (ECG) established and performed according to the characteristics of the drug during screening
6. From the date of first administration of the clinical trial drug to the date 7 days after the last administration, either you or your spouse agrees to exclude the possibility of pregnancy using medically appropriate contraception* and to not provide sperm or eggs
7. After hearing and fully understanding the full explanation for this clinical trial, the person who voluntarily decides to participate and agrees to comply with the precautions

Exclusion Criteria:

1. A person who has taken a drug metabolase-inducing and inhibiting drug, such as barbitals, within 30 days before the start of the test (the first day of administration), or who has taken a drug that may interfere with the main test within 10 days before the start of the test (the first day of administration)
2. Anyone who has consumed excessive smoking or caffeine or alcohol within one month prior to the first administration of the clinical trial drug (caffeine: > 5 cups/day, alcohol: male: > 21 cups/week, female: > 14 cups/week, tobacco: > 20 cigarettes/day), or who cannot stop smoking, caffeine and alcohol consumption during each hospitalization period
3. Where the tester determines that the drug may affect the test or the safety of the subject, if the drug is administered within 14 days before the first administration of the clinical trial drug or the general drug including health food and vitamin preparations within 7 days
4. A person who has participated in clinical trials (including biological equivalence tests) and administered experimental drugs within 6 months before the start of the trial (the first dosing date)
5. A person who has donated whole blood within 8 weeks before the start of the test (the first medication date) or donated ingredients within 2 weeks or received a blood transfusion within 4 weeks
6. A person who has a history of gastrointestinal diseases (Cron's disease, ulcerative colitis, etc.) or surgery (excluding simple appendectomy or hernia surgery) that may affect the absorption of drugs
7. A person who has a clinically significant disease or mental illness corresponding to the biliary tract, kidney, nervous system, immune system, respiratory system, urinary system, digestive system, endocrine system, blood and tumor, cardiovascular system, musculoskeletal system, or has the following manifestations or past history

   * Patients with type 1 diabetes, acute or chronic metabolic acidosis, and those with a history of ketoacidosis (including diabetic ketoacidosis), diabetic comas and total marriages, lactic acidosis, etc
   * Patients with severe heart failure or a history of heart failure (New York Heart Association (NYHA) classification 1,2,3,4 heart conditions)
   * liver dysfunction
   * Patients with moderate to severe renal impairment (eGFR <60 mL/min/1.73 m2)
   * Patients undergoing tests for intravenous administration of radioiodine contrast agents
   * Before and after 48 hours of surgery, patients with dehydration, severe infection or severe traumatic systemic disorder, acute myocardial infarction, sepsis
   * patients with malnutrition, starvation, weakness, pituitary dysfunction or adrenal insufficiency
   * As a result of performing a diagnostic test at the time of screening, a person who shows the following figures: AST or ALT or total bilirubin more than twice the upper limit of normal range
8. A person who has a history of clinically significant hypersensitivity reactions to other drugs or additives, including clinical trial drug
9. A person who has a history of drug abuse within one year of screening
10. In the case of women who are pregnant women and pregnant women who are pregnant or pregnant
11. A person who determines that the investigator is not suitable for participating in the clinical trial due to other reasons

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
AUCt of CKD-379 | Pre-dose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48 hours]
  Area under the concentration-time curve time zero to time
Cmax of CKD-379 | Pre-dose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48 hours
  Maximum plasma concentration of the drug

CONTACTS AND LOCATIONS:
Locations (1):
- Bumin Hospital, Gangseo-gu, Seoul, South Korea